CLINICAL TRIAL: NCT01519869
Title: Neoadjuvant Platinum-based Chemotherapy in Advanced Ovarian, Fallopian Tube, and Primary Peritoneal Carcinoma Trial Protocol
Brief Title: Trial of Chemotherapy in Ovarian, Fallopian Tube and Peritoneal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rachel Miller (Other)
Responsible Party: Sponsor-Investigator, Rachel Miller, Assistant Professor, Obstetrics and Gynecology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-GYN-098-MCC
Record Dates: First submitted 2012-01-18; First posted 2012-01-27 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-11

CONDITIONS: Primary Peritoneal Carcinoma; Ovarian Carcinoma; Fallopian Tube Carcinoma
Keywords: peritoneal; carcinoma; ovarian; fallopian tube; neoadjuvant chemotherapy; surgical debulking
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- neoadjuvant chemotherapy (Experimental): platinum-based neoadjuvant chemotherapy followed by interval surgical debulking with platinum-based adjuvant chemotherapy
  Interventions: Drug: neoadjuvant chemotherapy

INTERVENTIONS:
Drug: neoadjuvant chemotherapy — platinum-based neoadjuvant chemotherapy followed by interval surgical debulking with platinum-based adjuvant chemotherapy

SUMMARY:
This is a prospective study to evaluate the hypothesis that platinum-based neoadjuvant chemotherapy followed by interval surgical debulking with platinum-based adjuvant chemotherapy is associated with improved maximal surgical cytoreduction rates, comparable survival, decreased morbidity, and increased quality of life in patients with International Federation of Gynecologic Oncology stages IIIC and IV ovarian, primary peritoneal, or fallopian tube cancer when compared to historical controls and to evaluate the hypothesis that cancer induced inflammation is a predictor of poor prognosis and response to therapy in this group of ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven stage IIIC/IV epithelial ovarian cancer, primary peritoneal, fallopian tube carcinoma. If a core biopsy is not possible, fine-needle aspirate showing adenocarcinoma is acceptable in the setting of a pelvic mass and presence of metastasis outside the pelvis measuring at least 2 cm, regional lymph-node metastasis or proof of stage IV disease, and ratio of CA 125 to CEA greater than 25. If CA 125 to CEA ratio is 25 or lower, barium enema, gastroscopy, and mammography must be negative.
* Patients must have adequate:

  * Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1,500/μl, equivalent to Common Toxicity Criteria for Adverse Events v3.0(CTCAE) Grade 1. This ANC cannot have been induced or supported by granulocyte colony stimulating factors.
  * Platelets greater than or equal to 100,000/μl, CTCAE Grade 0-1. Renal function: Creatinine ≤1.5 x institutional upper limit of normal ULN), CTCAE Grade 1.
  * Hepatic function: Bilirubin ≤ 1.5 x ULN, CTCAE Grade 1.SGOT and alkaline phosphatase ≤ 2.5 x ULN, CTCAE Grade 1.
  * Neurologic function: Neuropathy (sensory and motor) less than or equal to CTCAE Grade 1.
  * Blood coagulation parameters: PT such that international normalized ratio (INR) is ≤ 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for management of venous thrombosis) and a PTT <1.2 x ULN.
* Patients must have a World Health Organization Performance Status ≤2.
* Patients must be a candidate for surgery.
* An approved informed consent must be signed by the patient.

Exclusion Criteria:

* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor are excluded. Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease.
* Patients with a known synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met: Stage not greater than IA, no more than superficial myometrial invasion, without vascular or lymphatic invasion, no poorly differentiated subtypes (including papillary serous, clear cell or other FIGO Grade 3 lesions).
* With the exception of non-melanoma skin cancer and other specific malignancies noted above, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last five years or whose previous cancer treatment contraindicates this therapy are excluded.
* Patients with acute hepatitis or active infection that requires parenteral antibiotics are excluded.
* Patients with World Health Organization Performance Status of 3 or 4.
* Patients who are pregnant or nursing.
* Patients under the age of 18.
* Patients with a pelvic mass of any size that is causing pain, or other subjective symptoms that are intolerable to the patient.
* Patients who are not candidates for interval surgical debulking secondary to significant medical comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Miller, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Chemotherapy
Started | 28
Completed | 27
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Achieve Maximal Surgical Debulking
Description: Percentage of patients that achieve maximal surgical debulking as defined by no gross residual disease following a Simon's 2-stage design.
Time Frame: 5 years
Population: Only twenty-five patients were evaluated for gross residual disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 25
Participants | 10

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Neoadjuvant Chemotherapy
All-Cause Mortality (participants affected / at risk) | 23/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 28/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemotherapy (N=28)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Allergic reaction (Immune system disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 6 (8)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 9 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 6 (10)
Diarrhea (Gastrointestinal disorders) | 5 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Fatigue (General disorders) | 15 (21)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6)
Lymphocyte count decreased (Investigations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (21)
Neutrophil count decreased (Investigations) | 11 (24)
Pain (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (20)
Platelet count decreased (Investigations) | 4 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Vomiting (Gastrointestinal disorders) | 7 (14)
Weight loss (Investigations) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
White blood cell decreased (Investigations) | 4 (8)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-11-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT01519869/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT01519869/ICF_001.pdf